CLINICAL TRIAL: NCT02102620
Title: Effectiveness of Triamcinolone Hexacetonide Intra-articular Injection in Interphalangeal Joints: a 12 Weeks Randomized Controlled Trial in Osteoarthritis Hand Patients
Brief Title: Corticosteroid Intra-articular Injection in Hands Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Natalia de Oliva Spolidoro Paschoal, Physician, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUSaoPauloRheum01
Record Dates: First submitted 2014-03-24; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Hands Osteoarthritis
Keywords: intra-articular injection; corticosteroid; osteoarthritis; Interphalangeal joint
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IAI triamcinolone hexacetonide (Experimental): Intra-articular injection with corticosteroid . The study group was called triamcinolone hexacetonide / lidocaine (TH / LD) and a control group, called lidocaine (LD).
  Patients in TH / LD group underwent corticosteroid IAI scheme in its most symptomatic interphalangeal (IP) joint composed with triamcinolone hexacetonide(TH) (20mg/ml) and 2% lidocaine without vasoconstrictor. The IAI was realized in the 0.3 ml dose (6mg) of TH for PIP and 0.2 ml (4 mg) of HT for DIP, always associated with 0.1 mL of 2% lidocaine. Paracetamol 750 mg / tablet were also used if required during the 12 weeks of follow-up (up to 03 tablets per day).
  Interventions: Drug: Intra-articular injection with corticosteroid
- IAI lidocaine (Placebo Comparator): Intra-articular injection with lidocaine. The LD group patients underwent IAI with only 2% lidocaine without vasoconstrictor in its most symptomatic IP joint. Paracetamol 750 mg / tablet were also used if required during the 12 weeks of follow-up (up to 03 tablets per day) . Both groups of patients underwent only one IAI in the most symptomatic joint and on a single occasion.
  Interventions: Drug: Intra-articular injection with lidocaine

INTERVENTIONS:
Drug: Intra-articular injection with corticosteroid — After rigorous antisepsis with alcoholic 0.5% chlorhexidine. Sterile insulin syringe BD ™ Ultra Fine needles 8 mm x 0.3 mm 30 G) was used in all patients. The anatomical place used for needle entry was located in the dorsal - lateral joint aspect. After the procedure, the injected joint was immobilized for 48 hours.
  Other Names: triancil
  Arms: IAI triamcinolone hexacetonide
Drug: Intra-articular injection with lidocaine — After rigorous antisepsis with alcoholic 0.5% chlorhexidine. Sterile insulin syringe BD ™ Ultra Fine needles 8 mm x 0.3 mm 30 G) was used in all patients. The anatomical place used for needle entry was located in the dorsal - lateral joint aspect. After the procedure, the injected joint was immobilized for 48 hours.
  Other Names: Xylestesin
  Arms: IAI lidocaine

SUMMARY:
Objective - to evaluate the effectiveness and tolerance of intra-articular injections (IAI) of hexacetonide triamcinolone (HT) for the treatment of osteoarthritis (OA) in interphalangeal joints.

Design:randomized, controlled, double-blinded study Materials and methods: sixty patients were randomized into: the TH / lidocaine (LD) group (n=30) who underwent IAI at the most symptomatic interphalangeal joint with HT (20mg/ml) and LD 2% or the LD group (n=30) who received IAI with just LD. Patients were assessed at baseline, 1, 4, 8 and 12 weeks by a blinded observer. The following parameters regarding the affected joint were assessed: pain at rest (VASr); pain at movement (VASm); pain (VAS) during the 48 hours after the procedure; swelling (VASs); goniometry; grip and pinch strength; hand function; treatment improvement; daily requirement of paracetamol and incidence and types of local side effects after the procedure.

DETAILED DESCRIPTION:
Background The aim of this study was to evaluate the effectiveness and tolerance of medium-term IAI of corticosteroids HT for the treatment of OA in proximal interphalangeal joints(PIP) or distal interphalangeal joints(DIP) joints on clinical and functional parameters.

Studies evaluating the effectiveness of intra-articular therapies in patients with hands OA are very heterogeneous, either by addressing different types of joints at the same time, for wearing unusual drugs, for failing to placebo groups , by using very soluble corticosteroid or not using corticosteroids.

Design A randomized, prospective, controlled, double-blinded, intention to treat study was performed.

Sample Patients were collected from the outpatient clinics of the Federal University of Sao Paulo, from August 2011 to August 2012. A total of 60 patients were randomized into two groups of 30 patients.

The patients had to fulfill the following inclusion criteria: diagnosis of PIP or DIP hands OA according to the American College of Rheumatology criteria, age greater than 40 years, and pain in at least one PIP or DIP hand joints between 3-8 cm on Visual Analog Scale for pain (VAS for pain at rest 0-10cm).

Patients with change in the corticosteroids or nonsteroidal antiinflammatory drug in the last thirty days; change in chondroprotective drugs in the last two months; IAI with corticosteroids in the studied joint in the last three months; any change in hand OA treatment in the last two months (rehabilitation, acupuncture and others); suspicion of local or systemic infection; hand x-ray suggesting another etiology of hand arthropathy (psoriatic arthritis, microcrystalline arthropathy, deposit disease) and severe coagulation disorder.

Intervention Patients were randomized into two groups. The study group was called hexacetonide triamcinolone / lidocaine (TH / LD) and a control group, called lidocaine (LD).

Patients in TH / LD group underwent treatment scheme in its most symptomatic interphalangeal (IP) joint composed of IAI with HT (20mg/ml) and 2% lidocaine without vasoconstrictor. The IAI was realized in the 0.3 ml dose (6mg) of HT for PIP and 0.2 ml (4 mg) of HT for DIP, always associated with 0.1 mL of 2% lidocaine. The LD group patients underwent IAI with only 2% lidocaine without vasoconstrictor in its most symptomatic IP joint. Paracetamol 750 mg / tablet were also used if required during the 12 weeks of follow-up (up to 03 tablets per day) for both groups. Both groups of patients underwent only one IAI in the most symptomatic joint and on a single occasion.

The procedures of the two groups were performed blindly by the same rheumatologist with 10 years of experience in interventional rheumatology after rigorous antisepsis with alcoholic 0.5% chlorhexidine. Sterile insulin syringe BD ™ Ultra Fine needles 8 mm x 0.3 mm 30 G) was used in all patients. The anatomical place used for needle entry was located in the dorsal - lateral joint aspect 14 (Figure 1). After the procedure, the injected joint was immobilized for 48 hours, in both groups.

Assessment All patients had their data reported in an evaluation form. The data collected were: age, sex, race, use of chondroprotective drugs, anti-inflammatory and / or analgesics drugs. Hands x-ray was performed in anteroposterior view for study inclusion. The measurement was done according to the method of Kellgren and Lawrence and used to evaluate homogeneity of the sample.

Five assessment evaluations were scheduled for a total of 12 weeks of follow-up. Patients were assessed at T0 (before intervention), T1, T4, T8 and T12 weeks after intervention. The assessment was carried out by a "blinded" assessor, trained in assessment instruments. This study was an intention to treat study. The last observation carried forward in case of discontinuation.

Clinical assessment

The following parameters were assessed in both groups:

* Visual analogue scale (VAS) for rest pain (VASr 0- 10cm);
* VAS for movement pain (VASm 0- 10cm);
* VAS for joint swelling (VASs 0- 10cm);
* Joint goniometry in flexion (degrees of range of motion);
* Analgesic consumption after the intervention (paracetamol daily average);
* Grip strength using Jamar® dynamometer (kgf) by obtaining the average of three attempts;
* Pinch strength using dynamometer Pinch Gauge (kgf) - by obtaining the average of three trials for the three types of pinches: tip, key and tripod 16;
* Hand function assessed by COCHIN questionnaire and the AUSCAN Index using the sub-scales pain, stiffness and hand function;
* Treatment improvement scale varying 5 points (much worse, worse , unchanged, little improvement and much improved);
* Side effects following the procedure (atrophy and / or cutaneous hypochromia and joint instability);
* Worsening of pain after IAI measured by VAS (post IAI VAS 0- 10cm) in 48 hours after the procedure (reported only at T1) in both groups.

Sample Size Using the VAS for pain as the primary study variable, considering a standard deviation equal to 1.5 points, based on previous work , and using the ANOVA for repeated measures as the statistical method for the calculation of the sample, with power of 90%, 5% significance and a detectable difference of 2.0 points on the VAS pain scale, measured 5 times over time into two independent groups, the investigators found a sample of 24 patients for each group. Considering a possible loss of up to 20% of patients over time, the investigators started the study with 30 patients in each group.

Randomization Patients were randomized using the MINITAB 14.0 software, with secret allocation guaranteed by opaque sealed envelopes. The responsible for the inclusion of these patients had no prior access to randomization list; it was responsible for verifying that the patient was within the inclusion and exclusion criteria of the study and after this procedure refer patients to the evaluators in another room, where medication was prepared.

Sample Blinding Only the responsible for the inclusion / exclusion of patients had access to which group the patient belonged, after enrollment. Evaluators and the responsible for the procedure had no access to such information. This blinding was relative impaired, since the volume used in the infiltration group TH / LD was substantially greater than that used in the LD group. However the responsible for the procedure was not responsible for the recruitment/allocation or evaluation of the sample. Regarding this essay the evaluators did not identify problems related to "blinding" during the study.

Statistical methods SPSS software version 17.0 (Chicago, IL) was used to perform statistical analysis. The descriptive statistics (mean, standard deviation, confidence interval 95%) was used to characterize the patients in groups. Continuous variables of the 2 groups at baseline were compared using the Student t test (for normally distributed variables) and the Mann-Whitney test (for variables with distribution not considered normal). Categorical variables were evaluated using the chi-square test.

To assess the response to intervention, analysis of variance (ANOVA) with repeated measures was used to intragroup and intergroup analysis over time.

This study was considered statistically significant if p values <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Hand OA
* Age over 40
* Visual analogic scale (VAS) for pain at rest between 3-8cm
* Signed informed consent term

Exclusion Criteria:

* Change in the use of oral corticosteroid or nonsteroidal antiinflammatory (NSAID) in the last 30 days
* Change in drugs for OA in the last two months
* IAI in this joints in the last three months
* Any change in treatment for OA in the hands in the last two months
* Suspicion of local and or systemic infection, and pregnancy
* Hands X-ray suggesting arthropathy of the interphalanges of other etiology
* Serious coagulation disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain Score on the Visual Analogue Scale (VAS) at 3 months | 0 -1-4-8 and 12 weeks
  To evaluate the improvement on pain measure by:VAS for rest pain (VASr 0- 10cm) and movement (VASm 0- 10cm) in each time

SECONDARY OUTCOMES:
Safety at 3 months | 0-1-4-8 and 12 weeks
  Side effects following the procedure (atrophy and / or cutaneous hypochromia and joint instability);

OTHER OUTCOMES:
Change from Baseline in Hand function at 3 months | 0-1-4-8 and 12 weeks
  Hand function assessed by COCHIN scale and the Australian/Canadian (AUSCAN)Osteoarthritis Hand Index using the sub-scales pain, stiffness and hand function.
Change from Baseline on Goniometry at 3 months | 0-1-4-8 and 12weeks
  Joint goniometry in flexion (degrees of range of motion)
Change from Baseline in Hand strength at 3 months | 0-1-4-8 and 12 weeks
  Grip strength using Jamar® dynamometer (kgf) by obtaining the average of three attempts; Pinch strength using dynamometer Pinch Gauge (kgf) - by obtaining the average of three trials for the three types of pinches: tip, key and tripod.
Change from Baseline in Analgesic consumption at 3 months | 0-1-4-8 and 12weeks
  Analgesic consumption after the intervention (paracetamol daily average).
VAS pain after procedure | 48 hours
  Worsening of pain after IAI measured by VAS (post IAI VAS 0- 10cm) in 48 hours after the procedure
Change from Baseline in Subjective analysis of improvement at 3 months | 1-4-8 and 12 weeks
  Treatment improvement scale varying 5 points (much worse, worse , unchanged, little improvement and much improved).

CONTACTS AND LOCATIONS:
Overall Officials: Natalia O Spolidoro Paschoal, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Spolidoro Paschoal Nde O, Natour J, Machado FS, de Oliveira HA, Furtado RN. Effectiveness of Triamcinolone Hexacetonide Intraarticular Injection in Interphalangeal Joints: A 12-week Randomized Controlled Trial in Patients with Hand Osteoarthritis. J Rheumatol. 2015 Oct;42(10):1869-77. doi: 10.3899/jrheum.140736. Epub 2015 Aug 1. PMID 26233501